CLINICAL TRIAL: NCT05768451
Title: Accurate Prediction of Breast Cancer and Axillary Lymph Node Metastasis Burden by Multi-modal Ultrasound-based Radiomics
Brief Title: Ultrasound Radiomics for Predicting Breast Cancer and Axillary Lymph Node Metastasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-YXZX-YX-08
Record Dates: First submitted 2022-12-05; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Axillary Lymph Node Metastasis
Keywords: breast cancer; multi-modal ultrasound; radiomics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- benign
  Interventions: Other: Ultrasonic image analysis
- malignant
  Interventions: Other: Ultrasonic image analysis

INTERVENTIONS:
Other: Ultrasonic image analysis — Preoperative conventional ultrasound (US), elastic ultrasound (UE) and contrast-enhanced ultrasound (CEUS) images were analyzed. Histopathological results were used as the gold standard. The cases were randomly divided into training set and test set with a ratio of 7:3. The US image, UE image and CEUS image of the maximum long-axis section of each lesion were selected, and the region of interest (ROI) of the lesion was manually delineated.

SUMMARY:
The project is proposed based on multimodal ultrasonic imaging omics building used for accurate prediction of the breast cancer and axillary lymph node metastasis load artificial intelligence forecasting model, this method can dig the hidden features of ultrasonic image is not visible to the naked eye, make up the subjectivity in the process of clinical doctors in diagnosis and treatment, provide accurate, objective basis for clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* patients who have not received breast puncture biopsy or neoadjuvant chemotherapy, etc. prior to ultrasonography;
* patients who are not allergic to the ultrasound contrast agent (SonoVue) and have signed an informed consent form for ultrasonography
* patients with breast tumors who have undergone surgical treatment at our hospital and have complete case histories.

Exclusion Criteria:

* patients with incomplete case data;
* cases with large breast masses that do not completely show the region of interest (ROI);
* patients who have undergone breast aspiration biopsy or other treatments such as neoadjuvant chemotherapy or endocrine therapy before ultrasound examination.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with breast tumors
Study Population: Patients with breast tumors seen in Nanjing Gulou Hospital in September 2018 and later and confirmed by histological pathology were selected, and all patients had complete preoperative US, UE and CEUS examination data.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of differential diagnosis between benign and malignant | 2022.12.15-2023.12.30
  ROC curve, sensitivity, specificity, accuracy, decision curve